CLINICAL TRIAL: NCT05846828
Title: Assesment of Cognitive Functions in Breastfed Preschool Children In Assiut Governorate, Egypt
Brief Title: Cognitive Functions in Breastfed Preschool Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Romany Eissa Atya Eissa, Principal Investigator, Assiut University
Other Study IDs: breastfeeding and IQ
Record Dates: First submitted 2023-03-31; First posted 2023-05-06 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Breast Feeding
Keywords: cognitive functions; IQ; Stanford binet test
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Stanford Binet IQ test — The Fourth Edition Stanford-Binet test which is based upon a four-factor model of intelligence, and its 15 subtests are partitioned into :
  1. Verbal ability.
  2. Abstract/Visual ability.
  3. Quantaitive potential.
  4. Short-Term Memory Scales

SUMMARY:
The current work aims to assess of the cognitive development in breastefed children and compare it with artificially fed children as well as the duration of breastfeeding.

DETAILED DESCRIPTION:
Breastfeeding provides nutritional and immunological benefits to infants and also prevents infections . Breastfeeding also has clear short-term benefits for child survival through reduction of morbidity and mortality from infectious diseases. Breastfeeding also has longterm benefits .Breastfeeding improves cognitive development and emotional interactions between the mother and infant .A previous meta-analysis of 20 studies that compared breastfeeding with formula-feeding reported that breastfeeding is associated with significantly improved cognitive development from infancy to adolescence .The results of a meta-analysis of these studies showed that breastfeeding was associated with an increase of 3•5 points (95% CI 1•9-5•0) on intelligence tests at childhood and adolescence. This beneficial effect of breastfeeding could be due to the presence of long-chain polyunsaturated fatty acids, such as arachidonic acid and docosahexaenoic acid in breast milk . Breastfed infants have higher concentrations of these fatty acids that are positively associated with brain development .

Child cognitive development is influenced by genetic and environmental factors . The child has a genetically determined potential for cognitive development. However environmental factors, such as adequate nutrition and the parents' ability to create a good and stimulating home environment may also have a positive influence on the child's cognitive development .Several studies have shown a positive correlation between breast feeding and cognitive development in children . In this study we measure the mental development of children by the use of Stanford binet intelligence test. It is a cognitive and intelligence test that is used diagnose developmental and intellectual deficiencies in young children .

Other risk factors affecting children's mental development should be taken in consideration like the mothers' age, educational level (lower than high school, high school diploma, college degree, university degree, and higher than a university degree), family income, job status (employed/unemployed), sex of infant, gestational age, and infant birth weight.

ELIGIBILITY:
Inclusion Criteria:

* Children more than 3 years and till age of 5 years that present to Assiut University Hospital with acute diseases.

Exclusion Criteria:

1. Children known to have chronic disease.
2. Chidren with History of birth anoxia, birth trauma, kernictrus, epilepsy, metabolic diseases.
3. Positive family history of mental retardation.

Ages: 3 Years to 5 Years | Sex: All
Age Groups: Child
Study Population: preschool children aged from 3 to 5 years
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
assess the cognitive development in breastefed children by the use of Stanford binet intelligence test and compare it with artificially fed children as well as the duration of breastfeeding. | Baseline
  In this study we measure the mental development of breast fed and artificailly fed preschool children by the use of Stanford binet intelligence test to prove that breastfed children have higher IQ than artificially fed chidren

CONTACTS AND LOCATIONS:
Overall Officials: Emad EL-Deen Mahmoud Hammad, prof, Principal Investigator — Assiut University; Amr Mohamed Kotb, lecturer, Principal Investigator — Assiut University

REFERENCES:
- [Background] Golding J, Rogers IS, Emmett PM. Association between breast feeding, child development and behaviour. Early Hum Dev. 1997 Oct 29;49 Suppl:S175-84. doi: 10.1016/s0378-3782(97)00062-5. PMID 9363425
- [Background] Fergusson DM, Beautrais AL, Silva PA. Breast-feeding and cognitive development in the first seven years of life. Soc Sci Med. 1982;16(19):1705-8. doi: 10.1016/0277-9536(82)90096-x. PMID 7178917
- [Background] Lee H, Park H, Ha E, Hong YC, Ha M, Park H, Kim BN, Lee B, Lee SJ, Lee KY, Kim JH, Jeong KS, Kim Y. Effect of Breastfeeding Duration on Cognitive Development in Infants: 3-Year Follow-up Study. J Korean Med Sci. 2016 Apr;31(4):579-84. doi: 10.3346/jkms.2016.31.4.579. Epub 2016 Feb 22. PMID 27051242